INSTITUTE/CENTER: National Cancer Institute
PRINCIPAL INVESTIGATOR: Azam Ghafoor, M.D.

STUDY NUMBER: 19C0127

**STUDY TITLE:** A Phase II Study of LMB-100 Followed by Pembrolizumab

in the Treatment of Adults with Mesothelin-Expressing Non-Squamous Non-Small Cell Lung Cancer

(NSCLC)

Cohort: Treatment after Progression

Consent Version: 12/04/2019

#### WHO DO YOU CONTACT ABOUT THIS STUDY?

**Study PI:** Azam Ghafoor, M.D.

Phone: 240-858-3289

Email: azam.ghafoor@nih.gov

## KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you to in making your decision about participating in this study. Additional information that may help you make a decision can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to take part in this study because after you began treatment with pembrolizumab on this study, it appears as if your tumors might have grown according to our scans. However, studies have shown that therapies such as pembrolizumab that target the immune system sometimes initially cause tumors to grow and then to later shrink. The initial growth is referred to as a tumor flare. Because of this feature of pembrolizumab, we cannot be certain after the first assessment that the study therapy is not working. Furthermore, your clinical condition has not gotten worse.

The purpose of this study is to continue treatment with pembrolizumab until we can be certain that the apparent increase in tumor size is not due to the tumor flare and is truly because your tumor is not responding to the pembrolizumab. It might take us several more cycles of therapy and several more scans to decide how to interpret your results.

Because it is standard practice to discontinue therapy at the first sign of tumor progression, we are asking your permission to continue with pembrolizumab therapy beyond this point.

# PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Protocol Number: [19C0127]


Refusing to do so will not affect your participation on this study. We would still want to keep in touch with you about your disease and any new therapies you might have started

Pembrolizumab (Keytruda®), is approved by the US Food and Drug Administration in the USA and some other countries for many cancers including NSCLC.

If you choose to remain on study therapy, you will continue to receive pembrolizumab as described in the study consent you signed when you enrolled and you will continue to have the same assessments (clinical and research). You will be required to continue on birth control as described in that consent.

In addition to the risks described in the first consent, continuing treatment as this point might lead you to miss out or cause a delay in your receiving alternative approaches as described below in the consent.

You are free to stop participating in the trial at any time. If you decide to stop, the study doctor may ask you to agree to certain tests to make sure it is safe for you to stop.

The remaining document will now describe more about the research study. This information should be considered before you make your choice. Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

If the individual being asked to participate in this research study is not able to give consent to be in this study, you are being asked to give permission for this person as their decision-maker. The term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research, throughout the remainder of this document.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

This is a research study.

We are asking you to continue on this research study because we would like to continue with pembrolizumab therapy beyond progression.

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Protocol Number: [19C0127]


Pembrolizumab (Keytruda®), is approved by the US Food and Drug Administration in the USA and some other countries for many cancers including NSCLC, but treatment beyond progression is not standard.

## WHAT WILL HAPPEN DURING THE STUDY?

If you choose to remain on study therapy, you will continue to receive pembrolizumab as described in the main study consent and you will continue to have the same assessments (clinical and research). You will be required to continue on birth control as described in the main consent.

# HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this study, your involvement will last for the rest of your life. The treatment portion of the study will last 2-3 years depending on whether you have a second course of pembrolizumab. You will be seen at least monthly during this time. After that, we will continue to follow you with scans and phone calls every 6-12 weeks as described in the standard consent.

# HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

Up to 23 people will be treated in this study at the NIH, however total 100 patients will be screened for the study.

#### WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

In addition to the risks described in the first consent, continuing treatment at this point might lead you to miss out on alternative approaches as described below.

## WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You might not benefit from being in this study.

The potential benefits are similar to what is described in the standard consent; however, as your tumor appears to have grown, it is more likely at this point than it was before that pembrolizumab may not have worked against your tumors.

# Are there any potential benefits to others that might result from the study?

In the future, other people might benefit from this study because what we learn in this study may eventually be used to treat others with your disease.

## WHAT OTHER OPTIONS ARE THERE FORYOU?

Instead of continuing pembrolizumab on this study, you have these options:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Protocol Number: [19C0127]


cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

There is no change in the criteria for stopping therapy and you will be allowed to discontinue therapy at any time you chose.

#### **DISCUSSION OF FINDINGS**

# New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

## Return of research results

There is no change from the first consent. Data will be returned as described in that document.

## EARLY WITHDRAWAL FROM THE STUDY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if your disease progress during treatment
- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you
- if you become pregnant
- if pembrolizumab become unavailable
- if you do not follow the study rules
- if the study is stopped for any reason

In this case, you will be informed of the reason therapy is being stopped.

After therapy is stopped we would like to see you for a safety visit 30 days and 90 days after your last dose.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you.

# WILL YOUR SPECIMENS OR DATA BE SAVED FOR USE IN OTHER RESEARCH STUDIES?

There is no change from the first consent. Specimens and data will be saved as described in that document.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Protocol Number: [19C0127]


# How Long Will Your Specimens and Data be Stored by the NIH?

Your specimens and data will be stored at the NIH indefinitely.

# Risks of Storage and Sharing of Specimens and Data

There is no change from the first consent. Specimens and data will be stored as described in that document.

# COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of my participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

The NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. Someone will work with you to provide more information.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment or related to care will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

# **CONFLICT OF INTEREST (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

The National Institutes of Health and the research team for this study have developed LMB-100 being used in this study. This means it is possible that the results of this study could lead to

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Protocol Number: [19C0127]


payments to NIH. By law, the government is required to share such payments with the employee inventors. You will not receive any money from the development of LMB-100.

# CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA) which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor (Center for Cancer Research)

When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

If we share your specimens or data with other researchers, in most circumstances we will remove your identifiers before sharing your specimens and data. You should be aware that there is a slight possibility that someone could figure out the information is about you.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Protocol Number: [19C0127]


## **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

# **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

## POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Protocol Number: [19C0127]


# PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Principal Investigator Azam Ghafoor, <u>azam.ghafoor@nih.gov</u> at 240-858-3289. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

## CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2)

Protocol Number: [19C0127]


# MEDICAL RECORD

# CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY

| <b>Adult Research Participant:</b> I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I consent to participate in this study. | | |
|---|---|---|
| Signature of Research Participant | Print Name of Research Participant | Date |
| <b>Legally Authorized Representative (LAR) for an Adult Unable to Consent:</b> I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I am legally authorized to make research decisions on behalf of the adult participant unable to consent and have the authority to provide consent to this study. As applicable, the information in the above consent was described to the adult participant unable to consent who agrees to participate in the study. | | |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Protocol Number: [19C0127]


IRB NUMBER: 19C0127

IRB APPROVAL DATE: 01/28/2020

# **MEDICAL RECORD**

CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY

| by the IRB for use as the basis of translation. | | |
|---|---|---|
| Witness: | | |
| Signature of Witness* | Print Name of Witness | Date |
| *NIH ADMINISTRATIVE SECTION TO INTERPRETER: | BE COMPLETED REGARDING T | THE USE OF AN |
| An interpreter, or other individual, who spectifies administration of informed consent and servalso serve as the witness. | | ~ ~ |
| An interpreter, or other individual, who speathe administration of informed consent but did no providing interpretive support is: | | ~ ~ |

Witness to the oral short-form consent process only: This section is only required if you are doing the oral short-consent process with a non-English speaking subject and this English consent form has been approved

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (2) Protocol Number: [19C0127]


IRB NUMBER: 19C0127

NIH) IRB APPROVAL DATE: 01/28/2020